CLINICAL TRIAL: NCT02198027
Title: Role of Peritubal Infiltration of 0.25% Bupivacaine in Percutaneous Nephrolithotomy (PCNL) in Postoperative Pain Control
Brief Title: Peritubal Infiltration of Bupivacaine in PCNL
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Indus Hospital and Health Network (Other)
Responsible Party: Principal Investigator, Zeeshan Arshad, Resident, Urology, Indus Hospital and Health Network
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: TIH-Urology-001; IRD_IRB_2014_01_002 (Other: IRD IRB)
Record Dates: First submitted 2014-07-21; First posted 2014-07-23 (Estimated); Last update posted 2014-09-23 (Estimated); Status verified 2014-09

CONDITIONS: Pain
Keywords: Percutaneous nephrolithotomy; postoperative analgesia; peritubal block; pain; Visual Analog Pain Scale
MeSH Terms: conditions — Pain | interventions — Bupivacaine; Saline Solution

STUDY DESIGN:
Who Masked: Participant, Care Provider, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Bupivacaine infiltration (Experimental): 10 ml of 0.25 % Bupivacaine
  Interventions: Drug: Bupivacaine
- Normal saline infiltration (Placebo Comparator): 10 ml of normal saline
  Interventions: Other: Normal saline infiltration

INTERVENTIONS:
Drug: Bupivacaine — 23 G spinal needle will be introduced along the nephrostomy tube for peri-tubal infiltration of 10 ml of 0.25 % Bupivacaine into renal capsule to skin.
  Arms: Bupivacaine infiltration
Other: Normal saline infiltration — 23 G spinal needle will be introduced along the nephrostomy tube for peri-tubal infiltration of 10 ml of normal saline into renal capsule to skin
  Other Names: normal saline
  Arms: Normal saline infiltration

SUMMARY:
Patients may feel significant pain at the surgery site after they wake up from the surgery. Usually pain is managed in the ward by giving strong pain medication that may slow down your mobilization and recovery process. Some recent work in other countries has shown that if investigator give patients an injection at the end of the operation, patients have less need for pain medication when they wake up. If investigator find that is also true in our population, then we can use this method as routine step after this operation to improve pain management and early mobilization of our patients

ELIGIBILITY:
Inclusion Criteria:

* Age 18-60 years of age
* Single PCNL track

Exclusion Criteria:

* Spinal Disc Prolapse
* Any previous renal surgery
* Complication secondary to PCNL

  * Hydrothorax that requires intervention
  * Pneumothorax
  * Massive hemorrhage that requires more than 1 U transfusion
  * Conversion to open procedure.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 68 (Estimated)
Dates: Start 2014-07; Primary Completion 2014-12 (Estimated); Study Completion 2014-12 (Estimated)

PRIMARY OUTCOMES:
Mean time for first demand of rescue analgesic | Release of the patient from the hospital or 24 hours (whichever comes first)
  Mean time for first demand defined as the difference in time between the first time rescue medications is given to patient in post-operatively and the time the infiltration took place intra-operatively

CONTACTS AND LOCATIONS:
Overall Officials: Zeeshan Arshad, MBBS, Principal Investigator — The Indus Hospital; Zafar Zaidi, MBBS, Study Director — The Indus Hospital
Locations (1):
- The Indus Hospital, Karachi, Sindh, Pakistan